CLINICAL TRIAL: NCT01623986
Title: Technical Correlation of a Noninvasive Estimation of Central Venous Pressure From the Mespere Venus 1000 System and the Inferior Vena Cava From Echocardiography, to Estimate Right Atrial Pressure
Brief Title: Correlation of Measurements From Mespere Venus 1000 System & Echocardiography to Estimate Right Atrial Pressure
Status: Completed | Type: Observational
Sponsor: Mespere Lifesciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MLS STP-9000010
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Patients Referred to St. Michael's Hospital Echocardiography Lab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- St. Michael's Hospital Patients: Patients who are referred to the St. Michael's Hospital echocardiography (ECHO) lab.
  Interventions: Device: Mespere Venus 1000 System; Device: Echocardiography machine

INTERVENTIONS:
Device: Mespere Venus 1000 System — An adhesive patch (connected to the Mespere Venus 1000 System) is placed on the neck of the subject, to determine if the CVP values displayed by the device correlates with right atrial pressure values obtained by echocardiography(standard clinical practice)
Device: Echocardiography machine — Use of ultrasound to estimate right atrial pressure from analyzing inferior vena cava (IVC).
  Other Names: ECHO machine

SUMMARY:
The purpose of this clinical study is to investigate if central venous pressure (CVP) measurements from the Mespere Venus 1000 System can be used for right atrial pressure (RAP) when estimating right ventricular systolic pressure (RVSP) in echocardiography labs.

DETAILED DESCRIPTION:
The non-invasive assessment of the pressure on the right side of your heart using an imaging machine called a Doppler echocardiography machine (also known as an ECHO machine) is a widely accepted technique and is used as a screening tool for pulmonary hypertension and heart failure. The pressure on this side of your heart reflects the pressure of the blood in your veins returning to your heart and the effectiveness of your heart to pump that blood to your lungs. The accuracy of this technique depends on making an accurate estimate of the pressure in the upper chamber (atrium) of the right side of your heart, known as your right atrial pressure (RAP). Right atrium pressure can be measured non-invasively by imaging of your heart using an echocardiography (aka ECHO) machine. But the technique depends on the skills of the sonographer (the person who operates the ECHO machine) and can take considerable time to complete.

In view of this limitation, a non-invasive technique that could be used to make the RAP measurements may be more reliable and/or faster than the current technique.

Mespere Lifesciences Inc. has developed a new non-invasive device that is expected to allow for a simple, rapid and reliable measurement of RAP. The device consists of a set of light sensors on a patch that is placed onto the surface of the patient's right side of the neck.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Patient referred to St. Michael's Hospital Echocardiography Lab
* Signed written and informed consent

Exclusion Criteria:

* Lack of patient consent
* Presence of known AV dialysis fistula
* Allergy to adhesive tape from Mespere Venus 1000 system
* Known central vein stenosis
* Unable to identify right external jugular vein
* Ongoing photodynamic therapy
* Assisted ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients referred to St. Michael's Hospital echocardiography lab
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Right atrial pressure (RAP) | 0-1 hour
  To determine if the RAP from the non-invasive Mespere Venus 1000 System correlates with the RAP from an echocardiography (ECHO) machine

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Ming Chow, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada